CLINICAL TRIAL: NCT05198908
Title: The Effect of Virtual Reality Glasse on Pain and Anxiety During Episiotomy Repair: Double-blind Randomized-Controlled Study
Brief Title: The Effect of Virtual Reality Glasse on Pain and Anxiety During Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KırklareliAS-5
Record Dates: First submitted 2021-12-18; First posted 2022-01-20 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Anxiety; Pain; Episiotomy Wound; Midwifery
Keywords: anxiety; pain; Episiotomy; Episiotomy wound; skin to contact; Midwifery
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR group (Experimental): VR (virtual reality glasse) group
  Interventions: Other: VR group
- skin to skin group (Experimental): skin to contact group
  Interventions: Other: Skin to skin group
- Control group-none (No Intervention): Women in this group will not be subjected to any treatment other than the routine hospital protocol. Before episiotomy repair, each woman is given superficial perineal anesthesia with a 4 ml ampoule of Jetocaine (ADEKA®, lidocaine HCl 40 mg/2 mL, epinephrine 0.025 mg/2 mL). This dose is repeated if necessary.

INTERVENTIONS:
Other: VR group — Women in this group will wear virtual reality glasses (15-20 minutes) until the episiotomy repair begins and ends. At the same time, the hospital protocol will be applied to this group.
  Before episiotomy repair, each woman is given superficial perineal anesthesia with a 4 ml ampoule of Jetocaine (ADEKA®, lidocaine HCl 40 mg/2 mL, epinephrine 0.025 mg/2 mL). This dose is repeated if necessary.
  Other Names: VR (virtual reality glasse) group
  Arms: VR group
Other: Skin to skin group — For women in this group, a warm sterile operating room towel will be placed on the newborn until the episiotomy repair begins and ends, so that her naked body remains on the mother's chest.At the same time, the hospital protocol will be applied to this group.
  Before episiotomy repair, each woman is given superficial perineal anesthesia with a 4 ml ampoule of Jetocaine (ADEKA®, lidocaine HCl 40 mg/2 mL, epinephrine 0.025 mg/2 mL). This dose is repeated if necessary.
  Other Names: Skin to contact group
  Arms: skin to skin group

SUMMARY:
Episiotomy is one of the common surgical operations that can cause anxiety in women and have side effects such as pain. Nerve blockades with analgesic effects such as lidocaine used during episiotomy repair or the use of tranquilizers and sleep-inducing drugs used to reduce anxiety during this procedure may have side effects. Nowadays, the trends towards non-medical methods (virtual reality glasses, praying, distraction, music therapy) in addition to medical methods during episiotomy repair are increasing due to the inevitable nature of these methods and the absence of side effects. In the study, it is stated that women will prefer non-medical methods (such as distraction or prayer) to alleviate pain or anxiety. It is important for midwives to have knowledge about these alternative methods (music therapy, virtual reality glasses, distraction, massage, acupressure, praying) to reduce the pain and anxiety that occurs during episiotomy repair. A new technology, virtual reality (VR), helps users connect to an environment that simulates reality, reducing pain by distracting them from the real world through computers or other devices. Although initially considered a technology only for the entertainment industry, its field of application has grown over the past decade to include various clinical areas such as pain management, physical rehabilitation, and psychiatric disorders. VR is suitable for clinical use and is a non-invasive and drug-free analgesic method. Its use in obstetrics is very new. Virtual reality glasses are recognized as a safe, inexpensive and effective non-pharmacological anxiolytic agent that allows for the reduction of regular pharmacological sedative doses due to their effect on anxiety and pain perception. Skin-to-skin contact is defined by the World Health Organization as the basic component of postnatal care. Skin-to-skin contact helps to reduce the pain felt during episiotomy repair in the mother and in the postpartum period. This research was planned to determine the effect of virtual reality glasses on pain and anxiety during episiotomy repair.

DETAILED DESCRIPTION:
Episiotomy is one of the common surgical operations that can cause anxiety in women and have side effects such as pain. Nerve blockades with analgesic effect such as lidocoin used during episiomy repair or the use of tranquilizers and sleep-inducing drugs used to reduce anxiety during this procedure may have side effects.This research was planned to determine the effect of virtual reality glasses and skin-to-skin contact application on pain and anxiety during episiotomy repair.This study is A prospective, double-blinded randomized controlled trial. Participants will randomized into VR, skin to contact, and control groups.Participants will be consisted of women over 20 years of age, 37-42. to be in the week of pregnancy, Singular pregnancy, being primiparous, Mediolateral episiotomy, Having a planned vaginal birth, Having a vertex presentation, Newborn APGAR score of 7 and above, Newborn weighing between 2-4 kg. In the selection of participants who meet the research criteria for the study, an introductory information form created by the researchers in the light of the literature will be used. Later, each method (VR,skin to contact and control group) will be evaluated for Visual Analog scale (VAS), State-Trait Anxiety Inventory (STAI).

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old,
* 37-42. to be in the week of pregnancy,
* Singular pregnancy, being primiparous,
* Mediolateral episiotomy,
* Having a planned vaginal birth,
* Having a vertex presentation,
* Newborn APGAR score of 7 and above,
* Newborn weighing between 2-4 kg,
* Signing the voluntary consent form, who has not used a non-pharmacological method before

Exclusion Criteria:

* Obstetric or non-obstetric complications
* Any obstetric complication or bleeding that requires urgent action,
* Using sedative drugs before and during episiotomy repair (except lidocaine applied in hospital routine),
* A condition that does not require episiotomy repair (small amounts of separation, etc.),
* Lacerations other than episiotomy (anal sphincter injury, 3rd or 4th degree laceration), episiotomies below 2 cm and above 4 cm,
* Instrument delivery (vacuum or forceps),
* Postpartum complications in the newborn,
* Chronic disease (Diabetes Mellus, thyroid, Hypertension),
* Regular drug use
* Having any problems that prevent communication (such as not knowing Turkish, hearing, speaking and understanding problems),
* Psychiatric treatment (Pharmacotherapy or psychotherapy).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Chance of pain felt during episiotomy repair | During study, an average of 1-1.5 hours
  The participants who met the inclusion criteria will included in the study. In practice, VAS will be administered separately to the women in the experimental groups and control group (pre-procedure, skin repair, immediately after skin repair, in the first hour after skin repair).
Chance of anxiety during episiotomy repair | Through study completion, an average of 1.5-2 hours
  The participants who met the inclusion criteria will included in the study.Participants in the experimental groups and control group will be followed for 1 hour in the delivery room after the episiotomy repair is completed.At the end of the follow-up, women who will be taken to the service will have the STAI scale filled.
Introductory Information Form | Approximately 5-10 hours (after hospitalization).
  This form, developed by the researchers in line with the literature, consists of 20 questions in total, including information about sociodemographic characteristics, medical and obstetric pregnancy history, and current pregnancy of the woman.
Visual Analog Scale (VAS) | Approximately 1-1.5 hours (during and after episiotomy repair)
  The scale was first developed and used by Bond and Pilowsky in 1966. The VAS is a 10 cm scale that expresses "painless" at one end and "worst pain" at the other. in VAS; 0 cm means "no pain", 0.5 cm - 3.0 cm means "mild pain", 3.5 cm - 6.5 cm means "moderate pain" and 7.0 cm - 10.0 cm means "severe pain". income.
State-Trait Anxiety Inventory (STAI) | Approximately 1.5-2 hours (after episiotomy repair)
  This scale, developed by Spielberg in 1973, consists of 20 questions. It is a 4-point Likert type scale (1=none, 4=very much). The lowest score that can be obtained from the scale is 20, and the highest score is 80. The higher the score, the higher the level of anxiety. The alpha value of the scale is 0.86-.92.33. Necessary permissions were obtained for the use of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Study Director — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No